CLINICAL TRIAL: NCT04670289
Title: A Phase 1, Single-Centre, Randomised, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability and Pharmacokinetics of Single Ascending Doses of TenoMiR Injections in Subjects With Lateral Epicondylitis
Brief Title: Safety, Tolerability, and Pharmacokinetics of Single Dose TenoMiR as a Treatment for Tennis Elbow
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Causeway Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CWT-TE1
Record Dates: First submitted 2020-11-26; First posted 2020-12-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Tennis Elbow
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: Prospective, Controlled, Randomised, Double Blind, Single Centre Trial
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): TenoMiR intralesional injection
  Interventions: Drug: TenoMiR (Low Dose); Drug: TenoMiR (Medium Dose); Drug: TenoMiR (High Dose)
- Placebo (Placebo Comparator): 0.9% saline intralesional injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TenoMiR (Low Dose) — Mimic of miR29a
  Other Names: CWT-001
  Arms: Treatment
Drug: TenoMiR (Medium Dose) — Mimic of miR29a
  Other Names: CWT-001
  Arms: Treatment
Drug: TenoMiR (High Dose) — Mimic of miR29a
  Other Names: CWT-001
  Arms: Treatment
Drug: Placebo — 0.9% saline
  Arms: Placebo

SUMMARY:
This study is testing a drug called TenoMiR that is being developed for the treatment of tennis elbow (lateral epicondylitis). The study drug is a new compound that works by improving the quality of the collagen which helps repair damage to the elbow. The study drug is being developed in the hope of providing a more reliable treatment than those currently available and can be given at the time of first diagnosis, so that recovery can begin as soon as possible.

DETAILED DESCRIPTION:
TenoMiR a chemically synthesised mimic of microRNA-29a (miR29a) which has improved stability, activity and cellular uptake while being non-immunogenic, has been created to restore miR29a levels back to pre-injury levels.

TenoMiR is unique in directly targeting the key changes in collagen production associated with tendinopathy. Unlike other therapies, TenoMiR has a well-defined mode-of-action that is supported by a wealth of scientific data. Moreover, treatment with TenoMiR does not require invasive biopsies and can be delivered at the point of initial diagnosis initiating recovery at the very earliest time.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a clinical diagnosis of lateral epicondylitis.
2. Aside from lateral epicondylitis, the subject is otherwise healthy as determined by a responsible physician, based on medical history, physical examinations, concomitant medication, vital signs, 12-lead ECGs and clinical laboratory evaluations. Laboratory values may be re-tested once at the discretion of the Investigator.
3. Subject's symptoms can be reproduced with resisted supination or wrist dorsiflexion (as confirmed by tenderness at lateral epicondyle and positive pick up back of chair sign).
4. Subject's symptoms have persisted for at least 6 weeks to 6 months, despite conservative treatment that includes 1 or combinations of:

   1. Physical therapy
   2. Splinting
   3. NSAIDs

Exclusion Criteria:

Subjects with any of the following will be excluded from study participation:

1. Subject has undergone previous corticosteroid injection therapy to the affected elbow in less than 6 months prior to enrolment.
2. Subjects unwilling or unable to discontinue use of pain medication (opiate or NSAID) from at least 1 week prior to Investigational Medicinal Product (IMP) administration.
3. Subject has received previous Platelet-Rich Plasma (PRP) injection to the affected elbow.
4. Subject uses or has recent use of medications known to affect the skeleton (e.g., glucocorticoid usage >5 mg/day, fluoroquinolone antibiotics).
5. Subject has undergone surgical intervention to the affected elbow for the treatment of lateral epicondylitis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AEs) as assessed by comparison of clinical laboratory abnormalities between TenoMiR versus placebo. | 14 days
  Comparison of clinical laboratory abnormalities between TenoMiR versus placebo as measured by blood chemistry, haematology, coagulation, serology and urinalysis.
Incidence of Treatment-Emergent Adverse Events (AEs) as assessed by comparison of changes in vital signs between TenoMiR versus placebo. | 14 days
  Comparison of changes in vital signs between TenoMiR versus placebo as measured by supine vital signs including pulse rate, blood pressure, respiration rate and oral temperature.
Incidence of Treatment-Emergent Adverse Events (AEs) as assessed by comparison of changes in 12 lead ECG parameters between TenoMiR versus placebo. | 14 days
  Comparison of changes in 12 lead ECG parameters as measured by Heart Rate and PR, RR, QRS, QT and QT intervals.
Incidence of Treatment-Emergent Adverse Events (AEs) as assessed by comparison of physical examination between TenoMiR versus placebo. | 14 days
  Comparison of changes in physical examination between TenoMiR versus placebo as measured by height, BMI, and body weight, and assessments of the head, eyes, ears, nose, throat, skin, thyroid, neurological, lungs, cardiovascular system, abdomen (liver and spleen), lymph nodes and extremities.
Incidence of Treatment-Emergent Adverse Events (AEs) as assessed by comparison of skin score assessment between TenoMiR versus placebo. | 14 days
  Comparison of changes in skin score assessment of injection site between TenoMiR versus placebo as measured by for erythema, pain, tenderness and swelling.

SECONDARY OUTCOMES:
Single dose pharmacokinetics (PK) of TenoMiR administration in subjects with lateral epicondylitis (Cmax). | 90 days
  Plasma PK by maximum drug plasma concentration (Cmax).
Single dose pharmacokinetics (PK) of TenoMiR administration in subjects with lateral epicondylitis (tmax). | 90 days
  Plasma PK by time to reach Cmax (tmax).
Single dose pharmacokinetics (PK) of TenoMiR administration in subjects with lateral epicondylitis (AUC). | 90 days
  Plasma PK by area under the plasma vs. concentration time curve (AUC).
Visual Analogue Score (VAS) pain score | 90 days
  Changes in pain score per group
Disabilities of the Arm, Shoulder, and Hand (Quick DASH) score | 90 days
  Changes in Quick DASH per group
American Shoulder and Elbow Surgeons Elbow (ASES-E) score | 90 days
  Changes in ASES-E per group
Patient Rated Tennis Elbow Evaluation (PRTEE) score | 90 days
  Changes in PRTEE per group
Ultrasound assessment | 90 days
  Change in analysis of focal hypoechoic areas within the tendon per group

CONTACTS AND LOCATIONS:
Locations (1):
- MAC Clinical Research, Manchester, United Kingdom